CLINICAL TRIAL: NCT06848335
Title: Improving Physical Activity Participation in Latinas With Mindfulness
Acronym: Seamos Activas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bess Marcus (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Lifespan/ The Miriam Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Bess Marcus, Professor of Behavioral and Social Sciences, Brown University
Organization: Brown University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL171195 (NIH); 1R01HL171195 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Inactivity; Inactivity/Low Levels of Exercise; Inactivity, Physical
Keywords: Physical Activity; Latinas; Spanish-Language; Text-Message; Exercise; Mindfulness
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remote Physical Activity Intervention (Experimental)
  Interventions: Behavioral: Remote Physical Activity Intervention
- Mindfulness Enhanced Remote Physical Activity Intervention (Active Comparator)
  Interventions: Behavioral: Mindfulness Enhanced Remote Physical Activity Intervention
- Attention Matched Enhanced Remote Physical Activity Intervention (Active Comparator)
  Interventions: Behavioral: Attention Matched Enhanced Remote PA intervention

INTERVENTIONS:
Behavioral: Remote Physical Activity Intervention — The intervention includes a Zoom goal setting session on PA at baseline and phone calls at week 1, and months 1, 2, 3, and 9 for new goal setting and to address questions and monitor progress on PA goals. Participants will receive mailings weekly in month 1, bi- weekly in months 2 and 3, and monthly in months 4 to 6, with maintenance doses in months 8 and 10. Mailings include motivation-matched physical activity manuals, tip sheets (on stretching, boredom, places to be active, etc.) and computer expert system-tailored PA feedback reports which draw from a bank of over 330 messages addressing psychosocial and environmental factors affecting PA. Participants receive one interactive text message on PA (goal setting and tips for increasing PA) daily for the first 6 months and weekly for months 7-12.
  Arms: Remote Physical Activity Intervention
Behavioral: Mindfulness Enhanced Remote Physical Activity Intervention — Women who do not meet the PA guidelines (60% based on our prior work), will be randomized to receive the Attention Matched Enhanced Remote PA intervention or Mindfulness enhanced remote Physical Activity intervention. The intervention includes a Zoom goal setting session on PA at baseline and phone calls at week 1, and months 1, 2, 3, and 9 for new goal setting and to address questions and monitor progress on PA goals. Participants will receive mailings weekly in month 1, bi- weekly in months 2 and 3, and monthly in months 4 to 6. In months 7-12, they will receive 4 monthly calls, 11 mailers and daily texts. In months 13-18, they will receive 1 call, weekly texts to self monitor daily PA and meeting goals. For the Mindfulness enhanced remote Physical Activity intervention participants will receive additional messaging and support to manage their stress through incorporating evidence based MBSR and mindful movement into their daily routine.
  Arms: Mindfulness Enhanced Remote Physical Activity Intervention
Behavioral: Attention Matched Enhanced Remote PA intervention — Women who do not meet the PA guidelines (60% based on our prior work), will be randomized to receive the Mindfulness enhanced remote Physical Activity intervention or the Attention Matched Enhanced Remote PA intervention as described here. The intervention includes a Zoom goal setting session on PA at baseline and phone calls at week 1, and months 1, 2, 3, and 9 for new goal setting and to address questions and monitor progress on PA goals. Participants will receive mailings weekly in month 1, bi- weekly in months 2 and 3, and monthly in months 4 to 6. In months 7-12, they will receive 4 monthly calls, 11 mailers and daily texts. In months 13-18, they will receive 1 call, weekly texts to self monitor daily PA and meeting goals.
  Arms: Attention Matched Enhanced Remote Physical Activity Intervention

SUMMARY:
In this study, the investigators are exploring how a mindfulness-based physical activity program can help improve exercise habits and overall health among 258 inactive Latina women aged 18 to 65. The study will be conducted entirely remotely over and 18 month period. During the first 6 months, all participants will receive an exercise program that has previously been tested by our research team. After 6 months, the investigators will check if participants are meeting the recommended exercise guidelines of at least 150 minutes/week of at least moderate intensity activity. Participants who meet the guidelines will continue with the successful exercise program for another 6 months. For participants who do not meet the guidelines (are exercising less than 150 minutes/week), they will receive one of two enhanced programs, which will be randomly assigned. One program offers additional physical activity support, and the other incorporates stress management through mindfulness techniques. For all participants, over 18 months, the investigators will track physical activity levels, stress, and heart health indicators.

DETAILED DESCRIPTION:
The current study is an innovative adaptive intervention tested on inactive Latinas aged 18-65 (n=258). During the initial 6 month phase, all participants will receive our evidence based physical activity (PA) intervention. At 6 months, participants who meet national PA guidelines (at least 150 mins/week of at least moderate intensity PA) will continue to receive the standard PA intervention for another 6 months. Participants who do not meet the PA guidelines, will be randomized to continue intensive PA counseling or receive attention matched PA counseling incorporating the most potent components from Mindfulness-Based Stress Reduction (MBSR) adapted for PA. Participants in all 3 arms will be followed and compared over 18 months. The investigators will also rigorously evaluate stress as a mechanism for meeting PA guidelines using multiple measures (objective and self-report), including using wearable technology and Ecological Momentary Assessment (EMA). Finally, heart health indicators will be collected to assess long term benefits of PA.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy (If asthma, controlled high blood pressure and/or controlled type II diabetes, may be able to participate with physician consent)
* Sedentary (defined as participating in MVPA for 60 minutes or less per week and engaging in muscle-strengthening exercise on less than 2 days per week)
* Hispanic or Latina (self-identified)
* Must be able to read and write in Spanish fluently
* 18 - 65 years of age
* Planning on living in the area for the next 18 months
* Own a cell phone capable of sending and receiving text messages
* Required to have reliable access to the Internet via a computer or mobile device
* Must be able to receive materials in the mail, either at your own home or at a mailbox

Exclusion Criteria:

* BMI greater than 45
* Not able to walk continuously for 30 minutes/limited ability to complete daily activity or ability to exercise
* Exercise is against advice of doctor
* Inability to walk independently
* Current or planned pregnancy in the next 12 months
* Heart disease/treatment
* Heart murmur
* Angina/chest pain or Angina/chest pain with exertion
* Palpitations
* Stroke/Transient Ischemic Attacks
* Peripheral Vascular Disease
* Diabetes that requires insulin
* Non-insulin dependent diabetes without physician approval to participate
* Chronic infectious disease- HIV, Hepatitis C but does not have doctor approval
* Chronic liver disease
* Cystic Fibrosis
* Abnormal EKG on last EKG performed
* Emphysema, Chronic bronchitis, Chronic Obstructive Pulmonary Disease
* Seizure in past year
* Surgery in past year on heart, lung, joint, orthopedic surgery
* Surgery pending in next year on lung, joint, orthopedic surgery
* Unusual/concerning shortness of breath
* Asthma (may be able to participate with physician consent)
* High blood pressure/high blood pressure medication (may be able to participate with physician consent)
* Use of Beta Blockers or medicines not approved by doctor.
* Abnormal Medical Stress Test in the last 12 months
* Musculoskeletal problems
* Fainting/dizziness more than 3 times in past year OR which interferes with daily activities OR causes loss of balance
* Cancer treatment in past 3 months
* Hospitalized for psychiatric disorder in past 3 years or suicidal
* Participation in prior Seamos Activas II study or participant in other research study about exercise currently or within the last 6 months ago

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 258 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-measured min/week MVPA | 12 and 18 Months (outcome timepoints)
  For the week prior to each assessment (baseline, 6, 12, 18-months), all participants will wear an Actigraph GT3X+ accelerometer, which measures movement and intensity of activity and has been validated against heart rate telemetry and total energy expenditure. Data will be used to generate a binary indicator of meeting national PA guidelines (at least 150 min/week MVPA) at each follow-up.

SECONDARY OUTCOMES:
Perceived Stress Scale(PSS) | Baseline, 6 months, 12 months, 18 months
  Measured using a 14-item Perceived Stress Scale(PSS), this self-report measure assesses general perceptions of demands in life exceeding one's capacities to manage them. This scale has shown good reliability and validity in past studies with Spanish speaking Latino participants. The scale score ranges from 0 to 56, with higher scores indicative of higher perceived stress.
Moment to moment self-reported stress evaluated via Ecological momentary assessment (EMA) | Baseline, 6, 9, 12 months
  Participants will be prompted daily (via the wake-up report and random prompts) to respond to : How stressed are you feeling right now? Response options are on a 7-point Likert scale ranging from 0=Not at all to 6=Extremely.

OTHER OUTCOMES:
Lipid Panel | Baseline, 6 months, 12 months, 18 months
  Heart health indicators will be collected at baseline and follow-ups (6, 12 and 18 months), including Total cholesterol, Triglycerides, HDL cholesterol and LDL cholesterol (all measured as mg/dl)
HbA1c | baseline, 6 months, 12 months, 18 months
  HbA1c will be collected at baseline, 6, 12, 18 months and is recorded as a percentage (mmol/mol).

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
All quantitative data produced in the course of the project will be preserved and shared upon reasonable request. Based on ethical considerations, only the following data produced in the course of the project will be preserved and shared: de-identified physical activity outcomes and questionnaire data.
Supporting Information: SAP
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication. The duration of preservation and sharing of the data will be a minimum of 7 years after the end of the funding period.
Access Criteria: Researchers will need to contact the study PI (Dr. Marcus)